CLINICAL TRIAL: NCT03588520
Title: Investigation Of The Utility Of Home Blood Pressure Measurements Towards Improving The Management Of Hypertension In Patients In Stage 3 And 4 Chronic Kidney Disease
Brief Title: Home Blood Pressure (HBP)-Guided Management of Hypertension in Stage 3-4 CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E. Champidou, Medical Doctor, Internal Medicine Specialist, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4475
Record Dates: First submitted 2018-06-30; First posted 2018-07-17 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Hypertension; Chronic Kidney Diseases
Keywords: Hypertension; Chronic Kidney Disease; Home Blood Pressure Monitoring; Blood Pressure Management; Masked Hypertension; White Coat Hypertension; Renal Insufficiency; Cardiovascular Risk
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Masked Hypertension; White Coat Hypertension; Renal Insufficiency | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home BP Monitoring Group (Experimental): Patients allocated to this group will receive a home blood pressure monitoring device and decisions to modify the hypertension treatment will be based on the results of the home blood pressure monitoring in accordance with the current guidelines of the European Society for Hypertension for the Treatment of Hypertension.
  Interventions: Diagnostic Test: Home Blood Pressure Monitoring
- Office BP Monitoring Group (No Intervention): Patients allocated to this group will act as controls. They will receive no home blood pressure monitoring device and decisions to modify the hypertension treatment will be based exclusively on blood pressure measurements in office visits.

INTERVENTIONS:
Diagnostic Test: Home Blood Pressure Monitoring — Patients randomly assigned to the HBP-guided management group will perform home BP monitoring for 7 days with the use of a validated self-inflating automatic oscillometric device (HEM 705 CP, Omron Healthcare). Home BP monitoring will be performed according to the currently available European Society of Hypertension guidelines at the baseline visit and will be repeated 1 week before the prespecified follow-up visits (at Month 1, Month 2 and Month 4). Patients randomly assigned to the control group will receive conventional management of hypertension based on office BP recordings obtained with the same BP monitor (HEM 705 CP, Omron Healthcare) during the same prespecified follow-up visits.
  Arms: Home BP Monitoring Group

SUMMARY:
It is estimated that over 25% of the world's population had hypertension in the year 2000 and that this proportion will reach 30% in the year 2025. With the introduction of the 2017 Guideline for High Blood Pressure in Adults from the American College of Cardiology and the American Heart Association Task Force on Clinical Practice Guidelines, the definition of hypertension became broader and as a result the prevalence is expected to further increase. On the other hand, it is estimated that around 10% of the world's population is affected by chronic kidney disease (CKD) with hypertension being both cause and complication of CKD.

It is obvious that hypertension and CKD are interconnected and are both major risk factors for cardiovascular disease (CVD). Hypertension results in increased CVD risk both directly, as an independent factor, and indirectly via its negative impact on renal function. In fact, the deterioration of the renal function is proportional to the degree of hypertension. On the other hand, the more advanced the CKD is, the more challenging the management of hypertension becomes, as patients with CKD present altered patterns of blood pressure (BP) during the day and, additionally, the prevalence of white coat and masked hypertension is significantly higher in this group of patients.

To date, hypertensive patients are treated according to the BP recordings that are obtained in the office (OBP) during routine patient visits, which leads to inaccurate estimates of the true burden of hypertension and also affects the efficacy of the therapeutic intervention. It has been suggested that self measured BP (HBP) is a more accurate estimate of the patients' daytime BP compared to the conventional office BP measurements. This has been already confirmed in studies regarding the general population and it has been suggested that the same applies to the patients with CKD. This study aims to check the validity of this hypothesis by comparing the effect of the HBP - guided management versus the conventional OBP - guided management on the 24 hour ambulatory BP monitoring of patients with uncontrolled hypertension and CKD stage 3 and 4.

DETAILED DESCRIPTION:
Hypertension among people with chronic kidney disease (CKD) is very common, difficult to diagnose and often poorly controlled. The identification and management of hypertension among patients with CKD is challenging, owing to the markedly altered patterns and rhythms of blood pressure (BP) during the 24-hour period (i.e., non-dipping status and nocturnal hypertension) and the high prevalence of white coat and masked hypertension in these individuals. Conventional BP recordings obtained in the office are reported to provide inaccurate estimates of the true BP burden assessed using out-of-office BP monitoring techniques. Self-measured BP by the patients themselves at home provides a more accurate estimate of the patient's daytime BP. Similarly to the general hypertensive population, clinical studies support the notion that among people with CKD, home BP monitoring offers several advantages over the conventional office BP recordings in diagnosing hypertension and estimating the associated cardiovascular and renal risk. Compared with office BP, home BP recordings exhibit closer association with indices of target-organ damage, such as left ventricular mass index and aortic pulse wave velocity (PWV). Moreover, compared with office BP, home BP recordings are stronger predictors of the rate of renal function decline over time and incident end-stage-renal-disease (ESRD) requiring dialysis. Importantly, home BP recordings were shown to carry stronger value relative to office BP in predicting the risk of all-cause and cardiovascular mortality.

The feasibility of performing repeated home BP monitoring over several days, weeks or months offers the ability to accurately assess alterations in BP levels and responses to antihypertensive therapy in the long-term. Consequently, several randomized controlled studies conducted in the general hypertensive population have provided evidence that home BP monitoring is a simple approach to guide the management of hypertension on a monthly basis. In a meta-analysis of 37 randomized controlled trials (incorporating data from 9,446 hypertensive patients), it was shown that compared with clinic BP-based hypertension management, home BP monitoring was associated with a significantly higher reduction in systolic BP [weighted mean difference (WMD): -2.63 mmHg; 95% Confidence Interval (CI): -4.24, -1.02] and in diastolic BP (WMD: -1.68 mmHg; 95% CI: -2.58, -0.79). Implementation of home BP monitoring as a tool to guide the management of hypertension was associated with more frequent reductions in the number of prescribed antihypertensive medications [relative risk (RR): 2.02; 95% CI: 1.32-3.11] and reduced the risk of therapeutic inertia, defined as unchanged antihypertensive regimen despite the presence of uncontrolled hypertension (RR: 0.82; 95% CI: 0.68-0.99).

In contrast to the accumulated evidence supporting the use of home BP (HBP)-guided management of hypertension in non-CKD populations, the only study to investigate the role of home BP monitoring as a tool to achieve BP targets in patients with CKD was a previous, small, randomized study enrolling 65 ESRD patients on maintenance hemodialysis. In this study the use of home BP monitoring for 6 months produced a significantly higher reduction in interdialytic ambulatory BP compared to conventional managements of hypertension based on routine pre-dialysis BP recordings (mean 24-hour BP at study-end: 135/76 versus 147/79 mmHg, p<0.05). Despite the fact that the use of home BP monitoring among people with hypertension and CKD is anticipated to overcome the barriers of white coat and masked hypertension effects and improve therapeutic inertia, there is still no solid evidence on the value of using this technique as a simple approach to improve BP control and maximize the associated benefits on regression of target-organ damage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or higher
* Stable CKD stage 3-4 (CKD-EPI estimated GFR: 15-60 ml/min/1.73m2)
* Treated or untreated uncontrolled hypertension, defined as office BP >140/90 mmHg for patients with diabetic or non-diabetic CKD and protein excretion <0.3 gr/day or office BP >130/80 mmHg for patients with diabetic or non-diabetic CKD and protein excretion ≥0.3 gr/day.22-24
* Patients must provide informed written consent

Exclusion Criteria:

* End-stage renal disease under hemodialysis or peritoneal dialysis
* Known secondary cause of hypertension (i.e., pheochromocytoma, primary aldosteronism, renovascular hypertension)
* Chronic atrial fibrillation
* Hospitalization for acute myocardial infarction, unstable angina or acute ischemic stroke within the 3 previous months
* Severe congestive heart failure stage III-IV according to New York Heart Association (NYHA) classification
* Body mass index (BMI) of >40 kg/m2
* History of malignancy or any other clinical condition associated with very poor prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-06-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Measurement | 4 months
  The difference in the change from baseline to 4 months in mean 24-hour ambulatory systolic, diastolic and mean BP between the HBP-guided management of hypertension and control groups.

SECONDARY OUTCOMES:
Office BP measurements | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the office systolic, diastolic and mean BP measurements
Hypertension Control Rates | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the hypertension control rates
Central Aortic BP | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the systolic, diastolic and mean central aortic BP
Carotid to femoral pulse wave velocity (cfPWV) | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the carotid to femoral Pulse Wave Velocity (cf PWV) and heart rate-adjusted augmentation index [AIx(75)]
Heart rate-corrected augmentation index AIx(75) | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in heart rate-adjusted augmentation index [AIx(75)]
Urinary protein excretion | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the urinary protein excretion
Urinary sodium excretion | 4 months
  The difference in the change from baseline to 4 months between HBP-guided management of hypertension and control groups in the Urinary protein excretion

OTHER OUTCOMES:
Secondary safety endpoint | 4 months
  The difference between the HBP-guided and conventional hypertension management groups in the occurrence of a composite of adverse events during the 4-month follow-up:
  1. symptomatic hypotension
  2. orthostatic hypotension
  3. acute renal injury
  4. progression of CKD to ESRD requiring dialysis
  5. cardiovascular death
  6. cardiovascular-related hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA University Hospital of Thessaloniki, Thessaloniki, Makedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarafidis PA, Li S, Chen SC, Collins AJ, Brown WW, Klag MJ, Bakris GL. Hypertension awareness, treatment, and control in chronic kidney disease. Am J Med. 2008 Apr;121(4):332-40. doi: 10.1016/j.amjmed.2007.11.025. PMID 18374693
- [Background] Sarafidis PA, Sharpe CC, Wood E, Blacklock R, Rumjon A, Al-Yassin A, Ariyanayagam R, Simmonds S, Fletcher-Rogers J, Vinen K. Prevalence, patterns of treatment, and control of hypertension in predialysis patients with chronic kidney disease. Nephron Clin Pract. 2012;120(3):c147-55. doi: 10.1159/000337571. Epub 2012 Jun 5. PMID 22678150
- [Background] Agarwal R, Pappas MK, Sinha AD. Masked Uncontrolled Hypertension in CKD. J Am Soc Nephrol. 2016 Mar;27(3):924-32. doi: 10.1681/ASN.2015030243. Epub 2015 Jul 10. PMID 26163421
- [Background] Cohen DL, Huan Y, Townsend RR. Home blood pressure monitoring in CKD. Am J Kidney Dis. 2014 May;63(5):835-42. doi: 10.1053/j.ajkd.2013.12.015. Epub 2014 Feb 12. PMID 24529535
- [Background] Gorostidi M, Sarafidis PA, de la Sierra A, Segura J, de la Cruz JJ, Banegas JR, Ruilope LM; Spanish ABPM Registry Investigators. Differences between office and 24-hour blood pressure control in hypertensive patients with CKD: A 5,693-patient cross-sectional analysis from Spain. Am J Kidney Dis. 2013 Aug;62(2):285-94. doi: 10.1053/j.ajkd.2013.03.025. Epub 2013 May 18. PMID 23689071
- [Background] Bangash F, Agarwal R. Masked hypertension and white-coat hypertension in chronic kidney disease: a meta-analysis. Clin J Am Soc Nephrol. 2009 Mar;4(3):656-64. doi: 10.2215/CJN.05391008. Epub 2009 Mar 4. PMID 19261815
- [Background] Parati G, Ochoa JE, Bilo G, Agarwal R, Covic A, Dekker FW, Fliser D, Heine GH, Jager KJ, Gargani L, Kanbay M, Mallamaci F, Massy Z, Ortiz A, Picano E, Rossignol P, Sarafidis P, Sicari R, Vanholder R, Wiecek A, London G, Zoccali C; European Renal and Cardiovascular Medicine (EURECA-m) working group of the European Renal Association-European Dialysis Transplantation Association (ERA-EDTA). Hypertension in Chronic Kidney Disease Part 2: Role of Ambulatory and Home Blood Pressure Monitoring for Assessing Alterations in Blood Pressure Variability and Blood Pressure Profiles. Hypertension. 2016 Jun;67(6):1102-10. doi: 10.1161/HYPERTENSIONAHA.115.06896. Epub 2016 May 2. No abstract available. PMID 27141057
- [Background] Parati G, Ochoa JE, Bilo G, Agarwal R, Covic A, Dekker FW, Fliser D, Heine GH, Jager KJ, Gargani L, Kanbay M, Mallamaci F, Massy Z, Ortiz A, Picano E, Rossignol P, Sarafidis P, Sicari R, Vanholder R, Wiecek A, London G, Zoccali C; European Renal and Cardiovascular Medicine (EURECA-m) working group of the European Renal Association-European Dialysis Transplantation Association (ERA-EDTA). Hypertension in Chronic Kidney Disease Part 1: Out-of-Office Blood Pressure Monitoring: Methods, Thresholds, and Patterns. Hypertension. 2016 Jun;67(6):1093-101. doi: 10.1161/HYPERTENSIONAHA.115.06895. Epub 2016 May 2. No abstract available. PMID 27141058
- [Background] Agarwal R. Arterial stiffness and its relationship to clinic and ambulatory blood pressure: a longitudinal study in non-dialysis chronic kidney disease. Nephrol Dial Transplant. 2017 Nov 1;32(11):1850-1856. doi: 10.1093/ndt/gfw281. PMID 27474747
- [Background] Agarwal R. Longitudinal Study of Left Ventricular Mass Growth: Comparative Study of Clinic and Ambulatory Systolic Blood Pressure in Chronic Kidney Disease. Hypertension. 2016 Apr;67(4):710-6. doi: 10.1161/HYPERTENSIONAHA.115.07052. Epub 2016 Feb 1. PMID 26831191
- [Background] Rave K, Bender R, Heise T, Sawicki PT. Value of blood pressure self-monitoring as a predictor of progression of diabetic nephropathy. J Hypertens. 1999 May;17(5):597-601. doi: 10.1097/00004872-199917050-00002. PMID 10403602
- [Background] Suzuki H, Nakamoto H, Okada H, Sugahara S, Kanno Y. Self-measured systolic blood pressure in the morning is a strong indicator of decline of renal function in hypertensive patients with non-diabetic chronic renal insufficiency. Clin Exp Hypertens. 2002 May;24(4):249-60. doi: 10.1081/ceh-120004229. PMID 12069356
- [Background] Agarwal R, Andersen MJ. Blood pressure recordings within and outside the clinic and cardiovascular events in chronic kidney disease. Am J Nephrol. 2006;26(5):503-10. doi: 10.1159/000097366. Epub 2006 Nov 22. PMID 17124383
- [Background] Minutolo R, Gabbai FB, Agarwal R, Chiodini P, Borrelli S, Bellizzi V, Nappi F, Stanzione G, Conte G, De Nicola L. Assessment of achieved clinic and ambulatory blood pressure recordings and outcomes during treatment in hypertensive patients with CKD: a multicenter prospective cohort study. Am J Kidney Dis. 2014 Nov;64(5):744-52. doi: 10.1053/j.ajkd.2014.06.014. Epub 2014 Jul 28. PMID 25082100
- [Background] Shimada K, Kario K, Kushiro T, Teramukai S, Zenimura N, Ishikawa Y, Okuda Y, Saito I. Prognostic significance of on-treatment home and clinic blood pressure for predicting cardiovascular events in hypertensive patients in the HONEST study. J Hypertens. 2016 Aug;34(8):1520-7. doi: 10.1097/HJH.0000000000000966. PMID 27310464
- [Background] Georgianos PI, Agarwal R. Epidemiology, diagnosis and management of hypertension among patients on chronic dialysis. Nat Rev Nephrol. 2016 Oct;12(10):636-47. doi: 10.1038/nrneph.2016.129. Epub 2016 Aug 30. PMID 27573731
- [Background] Agarwal R, Bills JE, Hecht TJ, Light RP. Role of home blood pressure monitoring in overcoming therapeutic inertia and improving hypertension control: a systematic review and meta-analysis. Hypertension. 2011 Jan;57(1):29-38. doi: 10.1161/HYPERTENSIONAHA.110.160911. Epub 2010 Nov 29. PMID 21115879
- [Background] Parati G, Stergiou GS, Asmar R, Bilo G, de Leeuw P, Imai Y, Kario K, Lurbe E, Manolis A, Mengden T, O'Brien E, Ohkubo T, Padfield P, Palatini P, Pickering T, Redon J, Revera M, Ruilope LM, Shennan A, Staessen JA, Tisler A, Waeber B, Zanchetti A, Mancia G; ESH Working Group on Blood Pressure Monitoring. European Society of Hypertension guidelines for blood pressure monitoring at home: a summary report of the Second International Consensus Conference on Home Blood Pressure Monitoring. J Hypertens. 2008 Aug;26(8):1505-26. doi: 10.1097/HJH.0b013e328308da66. PMID 18622223
- [Background] Stergiou GS, Bliziotis IA. Home blood pressure monitoring in the diagnosis and treatment of hypertension: a systematic review. Am J Hypertens. 2011 Feb;24(2):123-34. doi: 10.1038/ajh.2010.194. Epub 2010 Sep 9. PMID 20940712
- [Background] da Silva GV, de Barros S, Abensur H, Ortega KC, Mion D Jr; Cochrane Renal Group Prospective Trial Register: CRG060800146. Home blood pressure monitoring in blood pressure control among haemodialysis patients: an open randomized clinical trial. Nephrol Dial Transplant. 2009 Dec;24(12):3805-11. doi: 10.1093/ndt/gfp332. Epub 2009 Jul 8. PMID 19586971
- [Background] Hosseininasab M, Jahangard-Rafsanjani Z, Mohagheghi A, Sarayani A, Rashidian A, Javadi M, Ahmadvand A, Hadjibabaie M, Gholami K. Self-monitoring of blood pressure for improving adherence to antihypertensive medicines and blood pressure control: a randomized controlled trial. Am J Hypertens. 2014 Nov;27(11):1339-45. doi: 10.1093/ajh/hpu062. Epub 2014 Apr 26. PMID 24771706
- [Background] Botdorf J, Chaudhary K, Whaley-Connell A. Hypertension in Cardiovascular and Kidney Disease. Cardiorenal Med. 2011;1(3):183-192. doi: 10.1159/000329927. Epub 2011 Jul 30. PMID 22096454
- [Background] Judd E, Calhoun DA. Management of hypertension in CKD: beyond the guidelines. Adv Chronic Kidney Dis. 2015 Mar;22(2):116-22. doi: 10.1053/j.ackd.2014.12.001. PMID 25704348
- [Background] Gansevoort RT, Correa-Rotter R, Hemmelgarn BR, Jafar TH, Heerspink HJ, Mann JF, Matsushita K, Wen CP. Chronic kidney disease and cardiovascular risk: epidemiology, mechanisms, and prevention. Lancet. 2013 Jul 27;382(9889):339-52. doi: 10.1016/S0140-6736(13)60595-4. Epub 2013 May 31. PMID 23727170
- [Background] Bello AK, Levin A, Tonelli M, Okpechi IG, Feehally J, Harris D, Jindal K, Salako BL, Rateb A, Osman MA, Qarni B, Saad S, Lunney M, Wiebe N, Ye F, Johnson DW. Assessment of Global Kidney Health Care Status. JAMA. 2017 May 9;317(18):1864-1881. doi: 10.1001/jama.2017.4046. PMID 28430830
- [Background] Akobeng AK. Principles of evidence based medicine. Arch Dis Child. 2005 Aug;90(8):837-40. doi: 10.1136/adc.2005.071761. PMID 16040884
- [Background] Kabisch M, Ruckes C, Seibert-Grafe M, Blettner M. Randomized controlled trials: part 17 of a series on evaluation of scientific publications. Dtsch Arztebl Int. 2011 Sep;108(39):663-8. doi: 10.3238/arztebl.2011.0663. Epub 2011 Sep 30. PMID 22013494
- [Background] Levin KA. Study design VII. Randomised controlled trials. Evid Based Dent. 2007;8(1):22-3. doi: 10.1038/sj.ebd.6400473. PMID 17380181
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] DeLoach SS, Townsend RR. Vascular stiffness: its measurement and significance for epidemiologic and outcome studies. Clin J Am Soc Nephrol. 2008 Jan;3(1):184-92. doi: 10.2215/CJN.03340807. PMID 18178784
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Kidney Disease Outcomes Quality Initiative (K/DOQI). K/DOQI clinical practice guidelines on hypertension and antihypertensive agents in chronic kidney disease. Am J Kidney Dis. 2004 May;43(5 Suppl 1):S1-290. No abstract available. PMID 15114537
- [Background] Sarafidis PA, Ruilope LM. Aggressive blood pressure reduction and renin-angiotensin system blockade in chronic kidney disease: time for re-evaluation? Kidney Int. 2014 Mar;85(3):536-46. doi: 10.1038/ki.2013.355. Epub 2013 Sep 18. PMID 24048382
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Muntner P, Carey RM, Gidding S, Jones DW, Taler SJ, Wright JT Jr, Whelton PK. Potential US Population Impact of the 2017 ACC/AHA High Blood Pressure Guideline. Circulation. 2018 Jan 9;137(2):109-118. doi: 10.1161/CIRCULATIONAHA.117.032582. Epub 2017 Nov 13. PMID 29133599
- [Background] Levin A, Tonelli M, Bonventre J, Coresh J, Donner JA, Fogo AB, Fox CS, Gansevoort RT, Heerspink HJL, Jardine M, Kasiske B, Kottgen A, Kretzler M, Levey AS, Luyckx VA, Mehta R, Moe O, Obrador G, Pannu N, Parikh CR, Perkovic V, Pollock C, Stenvinkel P, Tuttle KR, Wheeler DC, Eckardt KU; ISN Global Kidney Health Summit participants. Global kidney health 2017 and beyond: a roadmap for closing gaps in care, research, and policy. Lancet. 2017 Oct 21;390(10105):1888-1917. doi: 10.1016/S0140-6736(17)30788-2. Epub 2017 Apr 20. PMID 28434650
- [Background] Kalaitzidis RG, Elisaf MS. Treatment of Hypertension in Chronic Kidney Disease. Curr Hypertens Rep. 2018 Jun 11;20(8):64. doi: 10.1007/s11906-018-0864-0. PMID 29892833